CLINICAL TRIAL: NCT02330848
Title: Walnut Ingestion in Adults at Risk for Diabetes: Effects on Body Composition, Diet Quality, and Cardiac Risk Measures
Acronym: Walnut3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-16
Record Dates: First submitted 2014-04-02; First posted 2015-01-05 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: Obesity; Walnuts; Endothelial Function; Adults at risk
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut Ad libitum diet (Active Comparator): Participants will be provided 392 grams of walnuts per week (56g or 2 oz/day) to include in their diet. Their calorie intake will not be subsequently monitored or regulated, and thus will be allowed to float ad libitum.
  Interventions: Dietary Supplement: Walnut Ad libitum diet
- Walnut Calorie Controlled (Active Comparator): The intervention group participants will meet with a registered dietitian and receive instructions and recipes for inclusion of 392 grams of walnuts per week (56g or 2 oz/day) in their meal plan. Participants will receive on-going instruction to preserve an isocaloric condition after the addition of walnuts. The study dietitian will customize dietary adjustments to make room for walnuts in the diet, while accommodating the priorities of each study participant. The general approach will emphasize general reduction in portion sizes; participants will also receive advice, based on baseline dietary intake analysis, of food eliminations that they might want to consider.
  Interventions: Dietary Supplement: Walnut Calorie controlled

INTERVENTIONS:
Dietary Supplement: Walnut Ad libitum diet — Participants will be provided 392 grams of walnuts per week (56g or 2 oz/day) to include in their diet. Their calorie intake will not be subsequently monitored or regulated, and thus will be allowed to float ad libitum
  Arms: Walnut Ad libitum diet
Dietary Supplement: Walnut Calorie controlled — The intervention group participants will meet with a registered dietitian and receive instructions and recipes for inclusion of 392 grams of walnuts per week (56g or 2 oz/day) in their meal plan for 6 months.
  Arms: Walnut Calorie Controlled

SUMMARY:
Proposed is a randomized, controlled, modified Latin square parallel design study with two treatment arms to examine walnut consumption effects on diet quality, body composition, and markers of cardiovascular risk in adults at risk for diabetes over a 6-month period. A modified crossover design (Latin square)27-29 will allow for both paired and unpaired analyses.

DETAILED DESCRIPTION:
Specific Aims

* To determine the effects of a walnut-included diet (with or without caloric intake adjustment) versus walnut-excluded diet on diet quality in adults at risk for diabetes. Specifically, to show that a walnut-included diet, as compared to a walnut-excluded diet will improve overall diet quality as measured by the Alternative Healthy Eating Index in adults at risk for diabetes.
* To determine the effects of a walnut-included diet (with or without caloric intake adjustment) versus walnut-excluded diet on body composition in adults at risk for diabetes. Specifically, to show that a walnut-included diet, as compared to a walnut-excluded diet for 6 months will improve body fat percentage in adults at risk for diabetes.
* To assess the effects of a walnut-included diet (with or without caloric intake adjustment) for a 6-month period on endothelial function, lipid panel levels, fasting glucose level, fasting insulin level and anthropometric measures in adults at risk for diabetes. Specifically, to show clinically meaningful improvement in endothelial function, lipid panel, fasting blood glucose, hemoglobin A1c (HbA1c), anthropometric measures and endothelial function with inclusion of walnuts in the diet in adults at risk for diabetes.

Hypotheses

* A walnut-included diet with or without dietary counseling to adjust caloric intake will improve diet quality in adults at risk for diabetes.
* A walnut-included diet for 6 months with or without dietary counseling to adjust caloric intake will improve body composition in adults at risk for diabetes.
* A walnut-included diet with or without dietary counseling to adjust caloric intake will improve lipid panel, fasting blood glucose, hemoglobin A1c, endothelial function and anthropometric measures in adults at risk for diabetes.
* Controlling calorie intake to keep it constant with the addition of walnuts to the diet will enhance the beneficial effects of walnut ingestion on diet quality, body composition, and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female age 25-75 years;
* Non-smoker;
* High risk for diabetes, defined as meeting at least one of the criteria listed below:

  a. Overweight with increased waist circumference; b.Pre-diabetes: fasting blood glucose >100mg/dL and <126mg/dL or HbA1C 5.7-6.4 % c. Metabolic syndrome, i.e. meet three out of five of the following criteria: i.Blood pressure >130/85 mmHg or currently taking antihypertensive medication; ii. Fasting plasma glucose (FPG) >100 mg/dL (6.1 mmol/L); iii.Serum triglycerides level (TG)>150 mg/dL (1.69 mmol/L); iv. High-density lipoprotein (HDL) cholesterol < 40 mg/dL (1.04 mmol/L) in men, and < 50 mg/dL (1.29 mmol/L) in women; v. Overweight (BMI ≥25kg/m²) with waist circumference of more than 40 inches (102 cm) for men and more than 35 inches (88 cm) for women.

Exclusion Criteria

* Allergy to walnuts or any other nuts;
* Anticipated inability to complete study protocol for any reason;
* Current eating disorder;
* Restricted diets by choice (i.e., vegetarian, vegan);
* Receiving pharmacotherapy for obesity, including appetite suppressant
* Unstable use of lipid-lowering, antihypertensive medications or aspirin (i.e. dose has changed in the three months prior to enrollment) or unwilling to refrain from taking medication for 12 hours prior to endothelial function scanning;
* Regular use of high doses of vitamin E (>400IU/day) or vitamin C (>500mg/day); fish oil, flaxseed oil, omega-3 fatty acid and fiber supplement unless welling to discontinue supplementation for the study duration.
* Use of insulin, glucose-sensitizing medication, vasoactive medication (including glucocorticoids, antineoplastic agents, psychoactive agents, or bronchodilators);
* Diagnosed diabetes;
* Diagnosed sleep apnea;
* Established cardiovascular disease (including symptomatic coronary artery disease (CAD), myocardial infarction, peripheral vascular disease, congestive heart failure, carotid stenosis);
* Coagulopathy, known bleeding diathesis, or history of clinically significant hemorrhage; current use of warfarin;
* Regular exercise defined as participation in moderate-intensity exercise > 150 minutes/week.
* Substance abuse (chronic alcoholism, other chemical dependency)
* Any unstable medical condition that would limit the ability of a subject to participate fully in the trial (e.g., cancer, AIDS, tuberculosis, psychotic disorder)
* Women who get Depo-Provera shots
* Women who are pregnant or lactating
* Women who are currently on hormone replacement therapy
* Substance abuse (chronic alcoholism, other chemical dependency)
* Any unstable medical condition that would limit the ability of a subject to participate fully in the trial (e.g., cancer, AIDS, tuberculosis, psychotic disorder)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Diet Quality assessed using the Alternative Healthy Eating Index (AHEI) | 6 months
  To help the study team track any variation in dietary pattern over the course of the study, all participants will be asked at five different time points to provide information on the foods and beverages that they consumed. A 3-day food diary record will be collected along with a one 24-hour recall using a web-based Automated Self-Administered 24-Hour Recall (ASA24) (available from the National Cancer Institute at http://riskfactor.cancer.gov/tools/instruments/asa24/) which will guide them through the process of completing the recall data. Diet quality will be assessed using the Alternative Healthy Eating Index (AHEI).

SECONDARY OUTCOMES:
Body Composition measured using bioelectrical impedance analysis and SC-240 Body Composition Analyzer | 6 months
  Body composition will be measured using bioelectrical impedance analysis, which uses the resistance of electrical flow through the body to estimate body fat. The Tanita SC-240 Body Composition Analyzer will be used to measure body composition. The SC-240 Body Composition Analyzer measures weight and calculates body fat% and total body water% in addition to BMI.
Endothelial Function (EF) Assessment using the brachial artery reactivity studies (BARS) methodology | 6 months
  The brachial artery reactivity studies (BARS) methodology employed is as described in the published, "Guidelines for Ultrasound Assessment of Endothelial-dependent Flow-mediated Vasodilation of the Brachial Artery." The measure of interest is flow-mediated dilatation of the brachial artery.
Anthropometric Measures | 6 months
  Body weight will be measured using a calibrated digital scale while height will be measured by using a calibrated stadiometer. Body mass index (BMI) will be calculated as weight (kg) divided by height in meters (m) squared. Waist circumference will be measured using guidelines of the National Obesity Expert Panel Report.
Lipid Profile | 6 months
  The lipid profile is determined as follows: Total cholesterol (Tchol), triglycerides (TRIG), and high-density lipoprotein (HDL) are obtained by direct measurements. Very-low-density lipoprotein (VLDL) and low-density-lipoprotein (LDL) are obtained by calculation: VLDL = TRIG/5; and LDL = Tchol - (VLDL + HDL). HDL:Tchol ratio will be used to evaluate the impact of walnuts on the lipid profile.
Fasting Blood Glucose | 6 months
HbA1C | 6 months
Physical Activity assessed by the International Physical Activity Questionnaire (IPAQ) | 6 months
  Physical activity will be assessed by the International Physical Activity Questionnaire (IPAQ). The IPAQ is a valid and reliable tool to assess physical activity in adults. It is a more comprehensive tool containing information on weekly activities in household and yard-work activities, occupational activity, transport, leisure time physical activity and sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: David L. Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Njike VY, Costales VC, Petraro P, Annam R, Yarandi N, Katz DL. The Resulting Variation in Nutrient Intake With the Inclusion of Walnuts in the Diets of Adults at Risk for Type 2 Diabetes: A Randomized, Controlled, Crossover Trial. Am J Health Promot. 2019 Mar;33(3):430-438. doi: 10.1177/0890117118791120. Epub 2018 Aug 1. PMID 30068215
- [Derived] Njike VY, Yarandi N, Petraro P, Ayettey RG, Treu JA, Katz DL. Inclusion of walnut in the diets of adults at risk for type 2 diabetes and their dietary pattern changes: a randomized, controlled, cross-over trial. BMJ Open Diabetes Res Care. 2016 Oct 19;4(1):e000293. doi: 10.1136/bmjdrc-2016-000293. eCollection 2016. PMID 27843557
- [Derived] Njike VY, Ayettey R, Petraro P, Treu JA, Katz DL. Walnut ingestion in adults at risk for diabetes: effects on body composition, diet quality, and cardiac risk measures. BMJ Open Diabetes Res Care. 2015 Oct 19;3(1):e000115. doi: 10.1136/bmjdrc-2015-000115. eCollection 2015. PMID 26688734